CLINICAL TRIAL: NCT06933147
Title: Comparative Effects of Resistance Training and Constrained Induced Movement Therapy on Upper Extremity Motor Recovery and Quality of Life in Sub-acute Stroke Patients
Brief Title: Resistance Training and Constrained Induced Movement Therapy on Upper Extremity Motor Recovery and Quality of Life in Sub-acute Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Hafiza Zoha Musharaf, Dr, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rec-UOL-/502/08/24
Record Dates: First submitted 2025-04-03; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Stroke
Keywords: Action Research Arm Test; Constraint-Induced Movement Therapy; Fugl-Meyer Assessment; Quality of Life; Resistance Training; Stroke Rehabilitation
MeSH Terms: conditions — Stroke | interventions — Constraint Induced Movement Therapy; Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Constraint-Induced Movement Therapy (CIMT) Group (Experimental): Participants in this group received Constraint-Induced Movement Therapy (CIMT) for 12 weeks. The unaffected upper limb was constrained for 6 hours per day using a mitt, and patients completed 3-hour daily sessions of task-specific functional training with the affected limb, 5 days per week. Exercises included grasping, stretching, pushing, button pressing, and fine motor tasks designed to improve upper limb function and daily activity performance. A home exercise plan was also provided.
  Interventions: Behavioral: Constraint-Induced Movement Therapy (CIMT)
- Resistance Training (RT) Group (Experimental): Participants in this group underwent Resistance Training (RT) focused on the affected upper extremity for 12 weeks. Exercises targeted shoulder, elbow, and wrist muscles using weight cuffs (½-1 kg) based on 1RM assessment. Each session included 3 sets of 8 reps for 4 different exercises, 5 days a week. The training started with 50% 1RM intensity for 4 weeks and progressed to 70% over the next 8 weeks. Sessions lasted 60 minutes and included rest intervals. A structured home exercise program was also provided.
  Interventions: Behavioral: Resistance Training (RT)

INTERVENTIONS:
Behavioral: Constraint-Induced Movement Therapy (CIMT) — This intervention involved constraining the unaffected upper limb for 6 hours per day and performing 3-hour intermittent daily sessions of functional task practice with the affected limb for 12 weeks, 5 days per week. Exercises included stretching, grasping, dexterity tasks, and functional activities like self-feeding and button pressing. The program used shaping techniques to increase task difficulty and improve motor recovery. A home exercise program was also prescribed for daily practice.
  Arms: Constraint-Induced Movement Therapy (CIMT) Group
Behavioral: Resistance Training (RT) — This intervention consisted of structured progressive resistance exercises targeting the affected upper limb muscles (shoulder, elbow, wrist) using weight cuffs (½-1 kg). Sessions were 60 minutes/day, 5 days/week, for 12 weeks. Intensity progressed from 50% to 70% of 1-repetition maximum (1RM) based on individual capacity. Exercises were performed in 3 sets of 8 repetitions for each muscle group, with 2-minute rest intervals. A home program included additional wrist and hand strengthening tasks.
  Arms: Resistance Training (RT) Group

SUMMARY:
This study explored two common rehabilitation strategies-Constraint-Induced Movement Therapy (CIMT) and Resistance Training (RT)-to help stroke survivors improve movement and function in their weaker arm. Stroke can often lead to reduced mobility in one arm, which affects a person's independence and quality of life. This randomized clinical trial involved 64 patients between the ages of 40 to 60 who had experienced a stroke and were in the sub-acute phase of recovery. Participants were randomly assigned to one of two groups: one group received CIMT and the other received RT. The CIMT group had their unaffected arm restrained for 6 hours per day and completed 3 hours of supervised exercises using the affected arm. The RT group participated in structured strength training using weights to target shoulder, elbow, and wrist muscles. Both groups were treated five days a week for 12 weeks. Throughout the study, researchers assessed participants using three tools: the Action Research Arm Test (ARAT) for arm function, the Fugl-Meyer Assessment (FMA) for motor recovery, and the Stroke-Specific Quality of Life Scale (SS-QOL) for overall well-being. These assessments were conducted at baseline, week 4, week 8, and week 12.

DETAILED DESCRIPTION:
This randomized clinical trial was designed to evaluate and compare the effects of two rehabilitation techniques-Constraint-Induced Movement Therapy (CIMT) and Resistance Training (RT)-on motor recovery and quality of life in patients recovering from sub-acute stroke. Stroke survivors commonly experience upper limb impairments that hinder their ability to perform activities of daily living (ADLs). Traditional therapy approaches often focus on general mobility, but targeted interventions like CIMT and RT have shown promise in enhancing specific motor functions and promoting neuroplasticity. A total of 64 stroke patients, aged 40-60 years, who had mild to moderate upper limb impairment were included. They were randomly assigned into two equal groups. Group A received CIMT, which involved constraining the unaffected arm for 6 hours daily and performing 3 hours of functional task-oriented training with the affected limb. Group B underwent RT, a progressive strengthening protocol that included concentric contractions of the shoulder, elbow, and wrist using weighted cuffs adjusted according to each patient's one-repetition maximum (1RM). Both groups received standard physiotherapy and were given home exercise programs. Patients were assessed using the Action Research Arm Test (ARAT), Fugl-Meyer Assessment (FMA), and Stroke-Specific Quality of Life Scale (SS-QOL) at four intervals: baseline, 4th week, 8th week, and 12th week. Data were analyzed using SPSS version 24. The study was ethically approved, and informed consent was obtained from all participants. It adhered to the ethical guidelines of the University of Lahore. Patients were assured of confidentiality, voluntary participation, and the right to withdraw at any point. No adverse effects were reported from either intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patient having age between 40-60 years
* Both gender were included
* Patient diagnosed with hemiparesis having grade 1 or 2 using Modified Ashworth Scale (MAS)
* Participant able to sit independently for 60 min
* Patients experiencing functional limitations in upper limb motor function

Exclusion Criteria:

* Participants with severe aphasia, severe shoulder pain affecting therapy or any comorbid condition that could limit UE function, visual or hearing impairment
* Uncontrolled pain or spasticity in the affected arm
* History of shoulder instability or major orthopedic surgery in the affected arm

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-03-19 (Actual); Study Completion 2025-04-02 (Actual)

PRIMARY OUTCOMES:
Action Research Arm Test (ARAT) | Baseline, Week 4, Week 8, and Week 12
  The ARAT is a standardized test used to assess upper extremity motor function. It evaluates grasp, grip, pinch, and gross arm movement using 19 items scored on a 4-point scale. Scores range from 0 to 57, with higher scores indicating better function.

SECONDARY OUTCOMES:
Fugl-Meyer Assessment (FMA) - Upper Extremity Section | Baseline, Week 4, Week 8, and Week 12
  The FMA is a widely used quantitative measure for assessing motor function, balance, and joint functioning in post-stroke patients. The upper extremity section scores range from 0 to 66, with higher scores indicating improved motor recovery.
Stroke-Specific Quality of Life Scale (SS-QOL) | Baseline, Week 4, Week 8, and Week 12
  The SS-QOL is a validated self-reported questionnaire measuring the quality of life in stroke survivors across 12 domains. It contains 49 items, scored on a 5-point Likert scale, with total scores ranging from 49 to 245 (higher scores indicate better quality of life).

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Lahore Teaching Hospital, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gracies JM, Pradines M, Ghedira M, Loche CM, Mardale V, Hennegrave C, Gault-Colas C, Audureau E, Hutin E, Baude M, Bayle N; Neurorestore Study Group. Guided Self-rehabilitation Contract vs conventional therapy in chronic stroke-induced hemiparesis: NEURORESTORE, a multicenter randomized controlled trial. BMC Neurol. 2019 Mar 12;19(1):39. doi: 10.1186/s12883-019-1257-y. PMID 30871480
- [Background] Lang CE, Strube MJ, Bland MD, Waddell KJ, Cherry-Allen KM, Nudo RJ, Dromerick AW, Birkenmeier RL. Dose response of task-specific upper limb training in people at least 6 months poststroke: A phase II, single-blind, randomized, controlled trial. Ann Neurol. 2016 Sep;80(3):342-54. doi: 10.1002/ana.24734. Epub 2016 Aug 16. PMID 27447365